CLINICAL TRIAL: NCT03853499
Title: Development of a Risk Score to Predict the Vacuum Extraction Failure
Acronym: FADS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2017/326
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-09

CONDITIONS: Vacuum Extraction
Keywords: Failure; Forceps Delivery; Cesarean Section; Affecting Fetus or Newborn; Vacuum Extraction
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful vacuum extraction: Patients for whom vacuum extraction was successful
  Interventions: Other: No intervention (observational study)
- Failed vacuum extraction: Patients who had an emergency caesarean section after failed vacuum extraction
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
Safe operative vaginal delivery requires a careful assessment of the clinical situation.

During the pushing efforts, the complexity of the delivery can lead to choose between an operative vaginal delivery attempt and a caesarean section straightaway. An emergency caesarean section for failed operative vaginal delivery is associated with a higher fetal and maternal morbidity, compared to a successful operative vaginal delivery and to a caesarean section straightaway.

The objective of this study was to develop a risk score of failed vacuum extraction leading to an emergency caesarean section.

This score could be an objective tool to help the obstetricians to choose between a vacuum extraction attempt and a caesarean section straightaway.

The investigators included patients who benefited from a vacuum extraction attempt in the Regional Teaching Hospital of Besançon (France) between January 2010 and December 2015. Patients were separated into two groups : the vacuum extraction failure group and the vacuum extraction success group.

The investigators selected maternal, fetal and labor characteristics which could influence success or failure of the vacuum extraction and compared them between the two groups.

The score was developed with the characteristics which significantly influence the vacuum extraction failure.

DETAILED DESCRIPTION:
Safe operative vaginal delivery requires a careful assessment of the clinical situation.

During the pushing efforts, the complexity of the delivery can lead to choose between an operative vaginal delivery attempt and a caesarean section straightaway. An emergency caesarean section for failed operative vaginal delivery is associated with a higher fetal and maternal morbidity, compared to a successful operative vaginal delivery and to a caesarean section straightaway.

The objective of this study was to develop a risk score of failed vacuum extraction leading to an emergency caesarean section.

This score could be an objective tool to help the obstetricians to choose between a vacuum extraction attempt and a caesarean section straightaway.

The investigators included patients who benefited from a vacuum extraction attempt in the Regional Teaching Hospital of Besançon (France) between January 2010 and December 2015. Patients were separated into two groups : the vacuum extraction failure group and the vacuum extraction success group.

The investigators selected maternal, fetal and labor characteristics which could influence success or failure of the vacuum extraction and compared them between the two groups.

The score was developed with the characteristics which significantly influence the vacuum extraction failure.

ELIGIBILITY:
Inclusion Criteria:

* delivery in the Regional Teaching Hospital of Besançon (France) between January 2010 and December 2015
* from 37 weeks of amenorrhea
* cephalic presentation
* epidural anesthesia
* vacuum extraction attempt (failure or success)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who delivered in the Regional Teaching Hospital of Besançon (France) between January 2010 and December 2015 and who met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1743 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Final mode of delivery | 1 year
  The final mode of delivery corresponds to :
  * a vacuum assisted vaginal delivery in case of successful vacuum extraction
  * an emergency caesarean section in case of failed vacuum extraction

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhoeven CJ, Nuij C, Janssen-Rolf CR, Schuit E, Bais JM, Oei SG, Mol BW. Predictors for failure of vacuum-assisted vaginal delivery: a case-control study. Eur J Obstet Gynecol Reprod Biol. 2016 May;200:29-34. doi: 10.1016/j.ejogrb.2016.02.008. Epub 2016 Mar 2. PMID 26967343
- [Background] Miot S, Riethmuller D, Deleplancque K, Teffaud O, Martin M, Maillet R, Schaal JP. [Cesarean section for failed vacuum extraction: risk factors and maternal and neonatal outcomes]. Gynecol Obstet Fertil. 2004 Jul-Aug;32(7-8):607-12. doi: 10.1016/j.gyobfe.2004.04.003. French. PMID 15450259
- [Background] Palatnik A, Grobman WA, Hellendag MG, Janetos TM, Gossett DR, Miller ES. Predictors of Failed Operative Vaginal Delivery in a Contemporary Obstetric Cohort. Obstet Gynecol. 2016 Mar;127(3):501-506. doi: 10.1097/AOG.0000000000001273. PMID 26855108
- [Background] Alexander JM, Leveno KJ, Hauth JC, Landon MB, Gilbert S, Spong CY, Varner MW, Caritis SN, Meis P, Wapner RJ, Sorokin Y, Miodovnik M, O'Sullivan MJ, Sibai BM, Langer O, Gabbe SG; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Failed operative vaginal delivery. Obstet Gynecol. 2009 Nov;114(5):1017-1022. doi: 10.1097/AOG.0b013e3181bbf3be. PMID 20168101
- [Background] Langeron A, Mercier G, Chauleur C, Varlet MN, Patural H, Lima S, Seffert P, Chene G. [Failed forceps extraction: risk factors and maternal and neonatal morbidity]. J Gynecol Obstet Biol Reprod (Paris). 2012 Jun;41(4):333-8. doi: 10.1016/j.jgyn.2011.11.001. Epub 2012 Jan 9. French. PMID 22227232
- [Background] Gopalani S, Bennett K, Critchlow C. Factors predictive of failed operative vaginal delivery. Am J Obstet Gynecol. 2004 Sep;191(3):896-902. doi: 10.1016/j.ajog.2004.05.073. PMID 15467561